CLINICAL TRIAL: NCT01051765
Title: Irinotecan Combined With Cisplatin as 1st Line Treatment for Esophageal Squamous Cell Cancer : a Single Center Prospective Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: zhang xiaodong, Peking University, School of Oncology, Department of GI oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-AEC1
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-05

CONDITIONS: Advanced Esophageal Squamous Carcinoma
MeSH Terms: interventions — Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan/cisplatin (Experimental): irinotecan 130mg/m2 d1 cisplatin: 30mg/m2, d1,d2 every three weeks
  Interventions: Drug: irinotecan/cisplatin

INTERVENTIONS:
Drug: irinotecan/cisplatin — irinotecan 130mg/m2 d1 cisplatin 30mg/m2, d1,d2 every 3 weeks

SUMMARY:
Irinotecan, as one new agent used in advanced esophageal carcinoma, has been shown to be effective and safe in western studies. Different with westerns, squamous carcinoma is the main pathological type in china patients. The investigators then initiated a prospective phase II clinical trial with irinotecan/cisplatin as the 1st line treatment in advanced esophageal carcinoma to observe the efficacy and safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age 18 to 70 years old
* Histologically confirmed esophageal squamous carcinoma, no prior palliative chemotherapy; recurrence from last adjuvant chemotherapy or adjuvant radiotherapy should be longer than 6 months; no prior treatment of irinotecan as adjuvant chemotherapy, total dose of cisplatin is less than 300mg/m2 if used in adjuvant chemotherapy
* Unresectable recurrent or metastatic disease
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Karnofsky performance status ≥70
* Life expectancy of ≥3 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
* Serum AKP < 2.5 times ULN (within 7 days before enrollment)
* Serum creatinine <1.0 times ULN (within 7 days before enrollment)
* Bilirubin level < 1.0 times ULN (within 7 days before enrollment)
* WBC>4,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl(within 7 days before enrollment)
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃；
* Good compliance

Exclusion Criteria:

* previous treatment of palliative chemotherapy or recurrence less than 6 months from time of last adjuvant chemo-/radiotherapy
* Known hypersensitivity to irinotecan
* Only with Brain or bone metastasis
* Tumor with length≥10cm, liver metastasis covers more than 50% of liver,or lung metastasis covers more than 25% of lung
* No measurable lesions, eg. pleural fluid and ascites
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months or
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 year

SECONDARY OUTCOMES:
PFS | 1year
response rate | 1.5 months
adverse events | 2 year
polymorphism of UGT1A | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Xiaodong, Beijing, Beijing Municipality, China